CLINICAL TRIAL: NCT04225364
Title: The Efficacy of Neoadjuvant PD-1 Plus Concurrent Chemotherapy for Stage II-IVA Operable Esophageal Squamous Cell Carcinoma：A Single Armed, Open-label, Multicentre, Clinical Trial
Brief Title: Efficacy of Neoadjuvant PD-1 Blockade Plus Chemotherapy for Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: BGI-Shenzhen (Industry); Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Liu, Clinical professor, Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIC-ESCC2019
Record Dates: First submitted 2019-12-23; First posted 2020-01-13 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Esophageal Squamous Cell Carcinoma; Immunotherapy
Keywords: neoadjuvant immunotherapy; Stage II-IVA; esophageal squamous cell carcinoma; ctDNA; neoadjuvant chemotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — camrelizumab; Paclitaxel; Injections; Cisplatin

STUDY DESIGN:
Intervention Model Description: Patients with II-IVA stage with pathologically diagnosed squamous cell lung carcinoma will be enrolled in this study. Camrelizumab plus chemotherapy will be administrated intravenously per 3 weeks at the dosage of 200mg. Contrast-CT evaluation and peripheral blood collected will be performed at pre-neoadjuvant therapy and pre-operation. 6 weeks after neoadjuvant therapy, participants who meet the indication will be assigned to operation. Another peripheral blood sample will be harvested 3-4 weeks after operation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- camrelizumab plus concurrent chemotherapy (Experimental): Neoadjuvant immunotherapy, PD-1, plus concurrent chemotherapy（albumin-bound paclitaxel + Cisplatin） will be applied to patients with operable esophageal squamous cell carcinoma before surgery.
  Interventions: Drug: camrelizumab; Drug: Paclitaxel for injection (albumin-bound); Drug: Cisplatin

INTERVENTIONS:
Drug: camrelizumab — Participants will receive camrelizumab, 200mg, intravenously over 30 - 60 minutes, day 1 of every 3 weeks for 6 weeks. Discontinuation will be considered due to toxicity, withdrawal of consent, or end of study. Every 3-week treatment period was considered to be a cycle.
  Other Names: SHR-1210
Drug: Paclitaxel for injection (albumin-bound) — Paclitaxel for injection (albumin-bound): 260mg/m2(in total), ivgtt d1, d8, q3w，for 2 cycle
  Other Names: paclitaxel
Drug: Cisplatin — 75mg/m2(in total), ivgtt d1-d3, q3w, for 2 cycles
  Other Names: CDDP

SUMMARY:
This study aims to evaluate the efficacy of Camrelizumab plus concurrent chemotherapy as neoadjuvant approach for patients with opearble esophageal squamous cell carcinoma. In addition, potential clinical utility of ctDNA in monitoring tumor burden and dynamics of tumor clonality during neoadjuvant immunotherapy will be assessed as well. At the same time, CD8 and PD-L1 will also be used as monitoring indicators.

DETAILED DESCRIPTION:
Immunotherapy improves clinical outcome of patients with advanced stage or metastatic esophageal squamous cell carcinoma (ESCC). In addition, superior effect of immunotherapy for esophageal squamous cell carcinoma was also reported recently. While, clinical application of ctDNA, PD-L1 and CD8 T cell monitoring in neoadjuvant immunotherapy for patients with esophageal squamous cell carcinoma is largely unknown. This trial will evaluate firstly the efficacy and the safety of Camrelizumab plus chemotherapy （albumin-bound paclitaxel plus cisplatin）as neoadjuvant approach. The evaluation indicators include pathological complete response rate (pCR) and objective imaging response rate after neoadjuvant therapy (ORR). ), 2-year progression-free survival (2y-PFS), postoperative progression-free survival (PFS), and overall survival (OS) after treatment. Objective response rate (ORR) based upon immune-Response Evaluation Criteria in Solid Tumors Version (RECIST v1.1). Major pathological response assessed by post-operational pathological review ctDNA efficacy will also be evaluated along with clinical management. Monitoring tumor burden, clonality as well as tumor heterogeneity evaluation will be correlated to radiological assessment and pathological findings.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ≥18 years, ≤70 years.
* Gastroscope/ultrasound gastroscopy biopsy, Histologically or cytologically confirmed esophageal squamous cell carcinoma. Clinically diagnosed as II-IVA esophageal squamous cell carcinoma (cT2N1-3M0/cT3N0-3M0/cT4N0-3M0).
* Non-Cervical Esophageal Cancer
* Previously received no systemic or topical treatment for esophageal cancer, at least one measurable lesion for neoadjuvant treatment imaging evaluation according to RECIST 1.1;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Estimated survival time ≥ 12 months;
* Subjects had no major organ dysfunction, and the investigators assessed thyroid, lung, liver, kidney function, and cardiac function as normal.
* Women of childbearing age must have taken reliable Contraception or have the negative predictive value of urine/ serum pregnancy test within 7 days prior to enrollment. They are also willing to use appropriate methods of contraception during the trial and 8 weeks after the last administration of the test drugs. For men, They must agree to use contraception or surgical sterilization during the trial and 8 weeks after the last administration of the test drug.
* Subjects voluntarily joined the study and signed informed consent. patients who accept blood sample collection at multiple time points. Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.

Exclusion Criteria:

* Have a history of gastrectomy or have surgical contraindications
* The investigator assessed that the patient had other serious illnesses that may affect follow-up and short-term survival;
* There are any active autoimmune diseases or a medical history of autoimmune (including, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, thyroid function Decreased. Subjects with vitiligo or adults who have had childhood asthma but have fully relieved without any intervention may be included. However, subjects who require bronchodilators for medical intervention cannot be included.)
* Cardiac clinical symptoms or diseases that are not well controlled, such as: a. Heart Failure NYHA > Class Ⅱ, b. unstable angina, c. myocardial infarction within 1 year; d. Clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention.
* Subjects with congenital or acquired immunodeficiency (such as HIV-infected), or active hepatitis (hepatitis B reference: HBsAg-positive, HBV DNA ≥ 2000 IU/ml or copy number ≥ 104/ml; hepatitis C reference: HCV antibody-positive.)
* Uncontrollable history of diabetes;
* Patients who have used other clinical trial study drugs within 4 weeks prior to the first dose.
* Severe allergic reactions to monoclonal antibodies or allergy to paclitaxel or human albumin.
* Peripheral blood neutrophil count is less than 1500/mm3
* Patients who have received or are undergoing other chemotherapy, radiation therapy or targeted therapy.
* According to the investigator's assessment, there are other factors that may lead to the termination of the study, such as other serious diseases (including mental illness) requiring combined treatment. Any other condition and social/psychological problems, etc., the investigator judged that the patient was not suitable for participation in the study.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Pathologic complete remission (PCR) | 4 weeks after surgery
  Primary tumor or lymph node surgery specimen pathological examination without residual tumor cell

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | At the end of Cycle 2 (each cycle is 21 days)
  Objective Response Rate Determine the tumor shrinkage rate, tumor boundary and the adhesion of tumor
2-year progression-free survival (PFS) | every 2 months (up to 24 months)
  From date of surgery until the date of first documented progression or date of death from any cause
Progression-free survival (PFS) | every 2 months (up to 24 months)
  From date of surgery until the date of first documented progression or date of death from any cause
Overall survival (OS) | every 2 months (up to 24 months)
  Defined from date of Signing ICF to date of first documentation of death from any cause or censored at the date of the last follow-up.

OTHER OUTCOMES:
safety of neoadjuvant PD-1 Blockade Plus Chemotherapy | Every 3 weeks (up to 3 months after surgery)
  Incidence of grade 3-5 adverse events [Safety and Tolerability]
Evaluation of molecular features and ctDNA changing in pre, per and post-treatment plasma | every 2 months (up to 12 months)
  All DNA samples were tested to calculate single nucleotide variants (SNV's), small insertions or deletions (Indels), copy number variations (CNV's), splice variations (SV's), gene fusions (GF's), tumor mutation burden (TMB) and micro-satellite instability (MSI) and others value by all enrolled. NGS (Next generation sequencing)-panel (688 genes) for monitoring on post-treatment residual disease in order to identify mechanisms of response. Measurement of different baseline ctDNA for their prognostic value.
Evaluation of Immunomicroenvironment changing in pre, per and post-treatment plasma | every 2 months (up to 12 months)
  the tumor immune microenvironment evaluated with multiplexed immunohistochemistry (mIHC), The evaluation of immune microenvironment uses the method of multiple immunofluorescence, through the detection of CD8, CD163, CD68, PD-1 and PD-L1 four bio-markers, determine the situation of related immune cells in the process and efficacy.
perioperative adverse events | Time to discharge or 30 days of in hospital stay whichever came first
  The participants were followed up daily and perioperative adverse events as defined by the American College of Surgeons National Quality Improvement Program. The participants were followed up until discharge or 30 days of in hospital stay and the secondary outcome measures entered into a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jun liu, Ph.D, M.D, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Jingpei Li, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Kang YK, Boku N, Satoh T, Ryu MH, Chao Y, Kato K, Chung HC, Chen JS, Muro K, Kang WK, Yeh KH, Yoshikawa T, Oh SC, Bai LY, Tamura T, Lee KW, Hamamoto Y, Kim JG, Chin K, Oh DY, Minashi K, Cho JY, Tsuda M, Chen LT. Nivolumab in patients with advanced gastric or gastro-oesophageal junction cancer refractory to, or intolerant of, at least two previous chemotherapy regimens (ONO-4538-12, ATTRACTION-2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Dec 2;390(10111):2461-2471. doi: 10.1016/S0140-6736(17)31827-5. Epub 2017 Oct 6. PMID 28993052
- [Background] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683
- [Background] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Lordick F, D'Journo XB, Cerfolio RJ, Korst RJ, Novoa NM, Swanson SJ, Brunelli A, Ismail M, Fernando HC, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J; AME Thoracic Surgery Collaborative Group. Neoadjuvant Chemoradiotherapy Followed by Surgery Versus Surgery Alone for Locally Advanced Squamous Cell Carcinoma of the Esophagus (NEOCRTEC5010): A Phase III Multicenter, Randomized, Open-Label Clinical Trial. J Clin Oncol. 2018 Sep 20;36(27):2796-2803. doi: 10.1200/JCO.2018.79.1483. Epub 2018 Aug 8. PMID 30089078